CLINICAL TRIAL: NCT02696304
Title: The Metabolic Syndrome Among Childhood Acute Leukemia Survivors: Physiopathological Analysis
Brief Title: The Metabolic Syndrome Among Leukemia Survivors: Physiopathological Analysis
Acronym: LEAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00170-49; 2015-05 (Other: APHM)
Record Dates: First submitted 2015-10-16; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2015-12

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TBI for childhood leukemia (Other): Patients with a metabolic syndrom who received TBI.
  Interventions: Other: Adipose tissu repartition; Other: Visceral and liver adipose tissue repartition; Other: Preadipocyte quantification and adipose tissue inflamation; Other: Inflamation blood markers quantification
- No TBI for childhood leukemia (Other): Patients with a metabolic syndrom without previousTBI
  Interventions: Other: Adipose tissu repartition; Other: Visceral and liver adipose tissue repartition; Other: Preadipocyte quantification and adipose tissue inflamation; Other: Inflamation blood markers quantification

INTERVENTIONS:
Other: Adipose tissu repartition — absorptiometry,
Other: Visceral and liver adipose tissue repartition — MRI,spectroscopy,
Other: Preadipocyte quantification and adipose tissue inflamation — biopsy
Other: Inflamation blood markers quantification — blood drawn,

SUMMARY:
Along with the improvement of childhood acute leukemia treatment, survival rates have increased. Therefore, the number of long term childhood leukemia survivors has increased progressively over the last decades. So, the assessment of long term health status in this population becomes very important. Many studies have shown an increased risk of life threatening late complications and early mortality. Cardiovascular morbidity and mortality are particularly frequent. Among these late complications, the metabolic syndrome (MS) is an important concern since it is associated with cardiovascular morbidity and mortality. The overall MS prevalence in the French prospective cohort of survivors of childhood acute leukemia was 9.2% and 18.6% in cases of total body irradiation (TBI) during the leukemia treatment. Since the median age at MS evaluation was 21 years, this prevalence was very high. Anyway, the MS pathophysiology in this population is still poorly understood. One of the most recent hypothesis about the MS mechanism is based on the adipose tissue inability to store fatty acids: when adipose tissue cannot expanse further to store excess nutriments then lipids accumulate in other tissues. This ectopic lipids accumulation can cause insulin resistance and MS.

The investigators hypothesized that the adipose tissue could be damaged by treatments received during childhood acute leukemia treatment (particularly TBI). This leads to morphological and functional abnormalities that could promote the insulin resistance and MS.

This ectopic adipose tissue contains less preadipocytes, which could impair its functional properties.

The primary endpoint of this study is to compare the morphological and functional characteristics of adipose tissue in patients with a MS who received or not TBI during childhood leukemia treatment . This comparison will focus on:

* The adipose tissue repartition and evaluation of the ectopic adipose tissue
* Fibrosis and inflammation of the adipose tissue
* Preadipocytes quantification

The secondary endpoint is to describe:

* for the whole cohort of included patients,
* the clinical and biological characteristics associated with the MS.
* Cardiovascular risk factors and nutritional statement
* Anthropometric measurements
* Detection of other endocrinal abnormalities possibly associated with the MS
* Analysis of inflammation blood markers and adipokines quantification.

DETAILED DESCRIPTION:
Enroled patients (both groups) will be evaluated for the following criteria. Then, a comparison between both groups will be performed.

1. Primary endpoint: the following factors will be studied, and compared between both groups (with or without TBI):

* Adipose tissue repartition using biphotonic absorptiometry and abdominal MRI
* Ectopic adipose tissue evaluation (visceral and hepatical) using MRI and proton spectroscopy
* Adipose tissue inflammation (using PCR array) : quantification of the following biomarkers: alpha TNF, IL6, IL1beta, IL10, MCP1, leptine and adiponectine
* Adipose tissue fibrosis (PCR array): quantification of the following markers of fibrosis: Col 1a1, Col 3a1, Col 6a1, Col 6a3, Tenascin C, Lumican, TGF beta
* Preadipocytes quantification in the adipose tissue (immunohistochemistery)

Concerning the secondary endpoints, the following points will be studied :

* Cardiovascular risk factors and nutritional statement
* Anthropometric measurements
* Other endocrinal abnormalities possibly associated with the MS
* Analysis of inflammation blood markers and adipokines quantification.

ELIGIBILITY:
Inclusion Criteria:

* Age superior or equal to 18 years
* Metabolic syndrome: at least 3 criteria among the following:

  1. Waist circumference ≥ 102 cm for male and ≥ 88 cm for female)
  2. High triglyceride level ≥ 150 mg/dl (1,7 mmol/l) or undergoing treatment for that affection
  3. Low HDL-Cholesterol < 40 mg/dl (1,03 mmol/l) for male ; < 50 mg/dl (1,3 mmol/l) for femal, or undergoing treatment for that affection
  4. Elevated blood pressure: systolic ≥ 130 mmHg and/or diastoloic ≥ 85 mmHg or undergoing treatment for that affection
  5. Elevated fasten glucose≥ 100 mg/dl or undergoing treatment for that affection
* Acute leukemia during childhood (under 18 years of age at the time of leukemia diagnosis)
* Informed consent obtained

Exclusion Criteria:

* pregnancy
* incomplete evaluation of metabolic syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percent of fat mass (Biphotonic absorptiometry) | 1 year
Evaluation of the amount of intra liver and pancreatic triglycerides (%) (proton spectroscopy, expressed as percent related to liver or pancreatic water content) | 1 year
Fibrosis and inflammation analyses of the adipose tissu : fibrosis and inflammation gene expression analyses by RQ-PCR | 1 year
Preadipocytes quantification in the adipose tissue by immunohistochemistery, expressed as percent of stroma vascular fraction of the adipose tissue | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM; Claire OUDIN, MD, Principal Investigator — AP-HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France